CLINICAL TRIAL: NCT04410523
Title: A 12-week, Multicenter, Randomized, Double-blind, Parallel-arm, Placebo-controlled Study to Assess the Efficacy and Safety of CSJ117, When Added to Existing Asthma Therapy in Patients ≥ 18 Years of Age With Severe Uncontrolled Asthma.
Brief Title: Study of Efficacy and Safety of CSJ117 in Patients With Severe Uncontrolled Asthma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Desicion
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCSJ117A12201C; 2019-004905-29 (EudraCT Number)
Record Dates: First submitted 2020-05-06; First posted 2020-06-01 (Actual); Results first posted 2023-08-07 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Asthma
Keywords: CSJ117; uncontrolled asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- CSJ117 0.5mg (Experimental): CSJ117 0.5 mg inhaled once daily
  Interventions: Drug: CSJ117; Drug: Placebo
- CSJ117 1mg (Experimental): CSJ117 1 mg inhaled once daily
  Interventions: Drug: CSJ117; Drug: Placebo
- CSJ117 2mg (Experimental): CSJ117 2 mg inhaled once daily
  Interventions: Drug: CSJ117; Drug: Placebo
- CSJ117 4mg (Experimental): CSJ117 4 mg inhaled once daily
  Interventions: Drug: CSJ117; Drug: Placebo
- CSJ117 8mg (Experimental): CSJ117 8 mg inhaled once daily
  Interventions: Drug: CSJ117; Drug: Placebo
- Placebo (Placebo Comparator): Placebo inhaled once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CSJ117 — CSJ117 inhaled once daily (in the morning) for 12 weeks. Delivered via Concept1 device.
  CSJ117 = inhaled monoclonal antibody fragment
  Arms: CSJ117 0.5mg; CSJ117 1mg; CSJ117 2mg; CSJ117 4mg; CSJ117 8mg
Drug: Placebo — Run-in period (all arms): Placebo inhaled once daily (in the morning) for 4 weeks. Placebo dosing extended to 8 weeks in case of asthma exacerbation or respiratory tract infection during this period.
  Treatment period (Placebo arm only): Placebo inhaled once daily (in the morning) for 12 weeks. Delivered via Concept1 device.

SUMMARY:
The purpose of this study is to determine the efficacy and safety of multiple CSJ117 doses (0.5; 1; 2; 4 and 8 mg) inhaled once daily compared with placebo, when added to standard-of-care (SoC) asthma therapy in adult patients with uncontrolled asthma with respect to change from baseline in FEV1 at the end of 12 weeks of treatment.

DETAILED DESCRIPTION:
This was a randomized, multicenter, multi-national, double-blind, placebo-controlled, parallel-arm study evaluating the effect of 5 dose levels of CSJ117 in adult subjects with inadequately controlled asthma despite medium to high dose inhaled corticosteroid (ICS) plus long-acting beta agonist (LABA).

Subjects were assigned to one of the following six treatment arms/groups in a ratio of 2:1:1:1:2:2:

* Placebo inhaled once daily
* CSJ117 0.5 mg inhaled once daily
* CSJ117 1.0 mg inhaled once daily
* CSJ117 2.0 mg inhaled once daily
* CSJ117 4.0 mg inhaled once daily
* CSJ117 8.0 mg inhaled once daily

The study included:

* A screening period of approximately 2 weeks
* A single blinded placebo run-in period of 4 weeks (extended to 8 weeks for subjects experiencing an asthma exacerbation or respiratory tract infection during the run-in period)
* A double blinded treatment period of 12 weeks
* A follow-up period of up to 12 weeks, study drug free, following the last dose of study treatment.

Patients who successfully completed 12 weeks of treatment in this study could be offered participation in the Safety Extension Study CCSJ117A12201E1 (NCT04946318).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed asthma
* Male and female patients aged ≥18 and ≤75 years
* Patients who have been treated with medium or high dose ICS plus LABA with up to 2 additional controllers
* Morning pre-BD FEV1 value of ≥ 40% and ≤ 85% of the predicted normal
* A positive reversibility test
* ACQ-5 score of ≥ 1.5 at screening and end of run-in visits.

Exclusion Criteria:

* Patients who have a cigarette smoking history of greater than 10 pack years or current smokers
* Pregnant or nursing (lactating) women
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using specified methods of contraception during dosing of study drug and until 12 weeks after last study drug treatment
* Patients with a history of immunodeficiency disease or hepatitis B, untreated and not cured hepatitis C or HIV.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-09-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (89):
- United States (19):
  - Novartis Investigative Site, Bakersfield, California
  - Novartis Investigative Site, Huntington Beach, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Mission Viejo, California
  - Novartis Investigative Site, San Jose, California
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Marietta, Georgia
  - Novartis Investigative Site, Bangor, Maine
  - Novartis Investigative Site, White Marsh, Maryland
  - Novartis Investigative Site, North Dartmouth, Massachusetts
  - Novartis Investigative Site, Columbia, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Boerne, Texas
  - Novartis Investigative Site, McKinney, Texas
- Argentina (12):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Mar del Plata, Buenos Aires
  - Novartis Investigative Site, Ranelagh, Partido de Berazate, Buenos Aires
  - Novartis Investigative Site, Concepción del Uruguay, Entre Ríos Province
  - Novartis Investigative Site, San Salvador, Entre Ríos Province
  - Novartis Investigative Site, Santa Fe, Rosario
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, CABA
  - Novartis Investigative Site, Mendoza
  - Novartis Investigative Site, Paraná
- Belgium (2):
  - Novartis Investigative Site, Erpent
  - Novartis Investigative Site, Liège
- Bulgaria (2):
  - Novartis Investigative Site, Rousse
  - Novartis Investigative Site, Stara Zagora
- Canada (6):
  - Novartis Investigative Site, Ajax, Ontario
  - Novartis Investigative Site, Burlington, Ontario
  - Novartis Investigative Site, Etobicoke, Ontario
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Trois-Rivières, Quebec
- Czechia (4):
  - Novartis Investigative Site, Teplice, CZE
  - Novartis Investigative Site, Jindřichův Hradec
  - Novartis Investigative Site, Lovosice
  - Novartis Investigative Site, Varnsdorf
- Germany (11):
  - Novartis Investigative Site, Peine, Lower Saxony
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Witten
- Guatemala (2):
  - Novartis Investigative Site, Guatemala City, GTM
  - Novartis Investigative Site, Guatemala City
- Hungary (5):
  - Novartis Investigative Site, Balassagyarmat
  - Novartis Investigative Site, Gödöllő
  - Novartis Investigative Site, Komárom
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szeged
- Japan (10):
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Kodaira, Tokyo
  - Novartis Investigative Site, Setagaya-Ku, Tokyo
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Toshima City, Tokyo
  - Novartis Investigative Site, Toshima Ku, Tokyo
  - Novartis Investigative Site, Osaka
- Latvia (3):
  - Novartis Investigative Site, Riga, LV
  - Novartis Investigative Site, Daugavpils
  - Novartis Investigative Site, Riga
- Philippines (3):
  - Novartis Investigative Site, Bulacan
  - Novartis Investigative Site, Iloilo City
  - Novartis Investigative Site, Manila
- Poland (4):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Poznan
- Russia (4):
  - Novartis Investigative Site, Izhevsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Ulyanovsk
- Slovakia (2):
  - Novartis Investigative Site, Levice
  - Novartis Investigative Site, Prešov

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- See also: Patient Lay Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1568

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 116 investigative sites in 15 countries.
Pre-assignment Details: The screening period of approximately 2 weeks began after the participants had provided written informed consent. There was a single blinded placebo run-in period of 4 weeks (extended to 8 weeks for subjects experiencing an asthma exacerbation or respiratory tract infection during the run-in period) before starting the double blinded treatment period.
Period: Overall Study
Arm/Group | CSJ117 0.5mg | CSJ117 1mg | CSJ117 2mg | CSJ117 4mg | CSJ117 8mg | Placebo
Started | 36 | 37 | 37 | 76 | 74 | 75
Completed | 32 | 32 | 35 | 69 | 71 | 65
Not Completed | 4 | 5 | 2 | 7 | 3 | 10
Not completed — Study terminated by sponsor | 1 | 3 | 2 | 6 | 3 | 4
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol deviation | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Subject decision | 2 | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CSJ117 0.5mg | CSJ117 1mg | CSJ117 2mg | CSJ117 4mg | CSJ117 8mg | Placebo | Total
Number analyzed (Participants) | 36 | 37 | 37 | 76 | 74 | 75 | 335
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (12.89) | 51.2 (12.09) | 51.4 (13.31) | 50.3 (12.80) | 52.7 (12.22) | 51.5 (13.46) | 51.3 (12.76)
Age, Customized [Count of Participants; unit: Participants]
  18 - <40 years | 9 | 6 | 8 | 16 | 10 | 19 | 68
  40 - <65 years | 23 | 26 | 23 | 50 | 50 | 41 | 213
  ≥65 years | 4 | 5 | 6 | 10 | 14 | 15 | 54
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 21 | 43 | 48 | 45 | 209
  Male | 9 | 12 | 16 | 33 | 26 | 30 | 126
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 8 | 8 | 7 | 17 | 16 | 17 | 73
  American Indian or Alaska Native | 1 | 3 | 0 | 1 | 1 | 3 | 9
  Black or African American | 1 | 0 | 0 | 2 | 5 | 2 | 10
  White | 26 | 26 | 30 | 56 | 52 | 53 | 243

OUTCOME MEASURES:

1. Primary Outcome: Average Change From Baseline in Pre-dose FEV1 at Week 8 and Week 12
Description: FEV1 (forced expiratory volume in one second) is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing.
  Pre-dose FEV1 is defined as average of the two FEV1 measurements taken at approximately 45 minutes and 15 minutes prior to dosing.
  The baseline pre-dose FEV1 value is defined as the average of the values taken approximately 2 hours 45 minutes and 2 hours 15 minutes prior to the first dose of double-blind treatment at Day 1.
  The least-squares means for change from baseline in pre-dose FEV1 averaged between Week 8 and Week 12 visits for each individual dose group were obtained from a linear mixed effects model for repeated measures (MMRM).
  A positive average change from baseline in pre-dose FEV1 is considered a favorable outcome.
Time Frame: Baseline, Weeks 8-12
Population: Full Analysis Set (FAS). The FAS included all participants to whom double-blind treatment had been assigned and who received at least one dose of double-blind treatment.
Measure: Least Squares Mean (Standard Error); unit: liters (L)
Arm/Group | CSJ117 0.5mg | CSJ117 1mg | CSJ117 2mg | CSJ117 4mg | CSJ117 8mg | Placebo
Number analyzed (Participants) | 36 | 37 | 37 | 76 | 74 | 75
liters (L) | 0.173 (0.0445) | 0.109 (0.0446) | 0.116 (0.0419) | 0.060 (0.0299) | 0.043 (0.0305) | 0.051 (0.0309)
Statistical Analysis 1: Comparison: CSJ117 0.5mg vs Placebo; Test type: Superiority; p = 0.025, MMRM; Least Squares mean = 0.122, 95% CI 2-sided [0.016 to 0.229], Standard Error of Mean 0.0541 — Treatment difference (CSJ117-placebo)
Statistical Analysis 2: Comparison: CSJ117 1mg vs Placebo; Test type: Superiority; p = 0.286, MMRM; Least Squares mean = 0.058, 95% CI 2-sided [-0.049 to 0.165], Standard Error of Mean 0.0542 — Treatment difference (CCSJ117-placebo)
Statistical Analysis 3: Comparison: CSJ117 2mg vs Placebo; Test type: Superiority; p = 0.212, MMRM; Least Squares mean = 0.065, 95% CI 2-sided [-0.037 to 0.168], Standard Error of Mean 0.0521 — Treatment difference (CCSJ117-placebo)
Statistical Analysis 4: Comparison: CSJ117 4mg vs Placebo; Test type: Superiority; p = 0.831, MMRM; Least Squares mean = 0.009, 95% CI 2-sided [-0.076 to 0.094], Standard Error of Mean 0.0430 — Treatment difference (CCSJ117-placebo)
Statistical Analysis 5: Comparison: CSJ117 8mg vs Placebo; Test type: Superiority; p = 0.852, MMRM; Least Squares mean = -0.008, 95% CI 2-sided [-0.094 to 0.077], Standard Error of Mean 0.0434 — Treatment difference (CCSJ117-placebo)

2. Secondary Outcome: Average Change From Baseline in FeNO at Week 8 and Week 12
Description: Fractional exhaled Nitric Oxide (FeNO) pre-dose measurements were done at the investigational sites prior to spirometry assessments. FeNO is defined as the mean of two serial measurements. The measurement of exhaled nitric oxide is widely accepted as a non-invasive marker of airway inflammation (inflammation leads to elevation of FeNO).
  The baseline FeNO pre-dose measurements were taken at the end of the run-in period.
  The least-squares means for change from baseline in FeNO averaged between Week 8 and Week 12 visits for each individual dose group were obtained from a linear mixed effects model for repeated measures (MMRM).
  A negative average change from baseline in FeNO is considered a favorable outcome.
Time Frame: Baseline, Weeks 8-12
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: parts per billion (ppb)
Arm/Group | CSJ117 0.5mg | CSJ117 1mg | CSJ117 2mg | CSJ117 4mg | CSJ117 8mg | Placebo
Number analyzed (Participants) | 36 | 37 | 37 | 76 | 74 | 75
parts per billion (ppb) | -2.869 (1.9670) | -5.299 (1.9872) | -4.190 (1.8760) | -1.587 (1.3312) | -0.208 (1.3248) | -1.301 (1.3142)
Statistical Analysis 1: Comparison: CSJ117 0.5mg vs Placebo; Test type: Superiority; p = 0.508, MMRM; Least Squares mean = -1.568, 95% CI 2-sided [-6.219 to 3.083], Standard Error of Mean 2.3630 — Treatment difference (CSJ117-placebo)
Statistical Analysis 2: Comparison: CSJ117 1mg vs Placebo; Test type: Superiority; p = 0.095, MMRM; Least Squares mean = -3.998, 95% CI 2-sided [-8.691 to 0.695], Standard Error of Mean 2.3840 — Treatment difference (CCSJ117-placebo)
Statistical Analysis 3: Comparison: CSJ117 2mg vs Placebo; Test type: Superiority; p = 0.209, MMRM; Least Squares mean = -2.889, 95% CI 2-sided [-7.405 to 1.627], Standard Error of Mean 2.2943 — Treatment difference (CCSJ117-placebo)
Statistical Analysis 4: Comparison: CSJ117 4mg vs Placebo; Test type: Superiority; p = 0.878, MMRM; Least Squares mean = -0.287, 95% CI 2-sided [-3.971 to 3.398], Standard Error of Mean 1.8718 — Treatment difference (CCSJ117-placebo)
Statistical Analysis 5: Comparison: CSJ117 8mg vs Placebo; Test type: Superiority; p = 0.558, MMRM; Least Squares mean = 1.093, 95% CI 2-sided [-2.578 to 4.765], Standard Error of Mean 1.8652 — Treatment difference (CCSJ117-placebo)

3. Secondary Outcome: Change From Baseline in Morning PEF at Week 12
Description: PEF (Peak Expiratory Flow) is a person's maximum speed of expiration. All participants were instructed to record PEF twice daily before taking any medication using an electronic peak expiratory flow device (eDiary/ePEF), once in the morning and once approximately 12 hours later in the evening at home. At each timepoint, the participant was instructed to perform 3 consecutive manoeuvres within 10 minutes. These PEF values were captured in the eDiary/ePEF.
  Mean morning and evening PEF values were calculated by weekly intervals. The baseline values of PEF were the mean values in the run-in period. A positive change from baseline in PEF is considered a favorable outcome.
Time Frame: Baseline, Week 12
Population: Participants in the Full Analysis Set with a valid measurement for the outcome measure
Measure: Mean (Standard Deviation); unit: liters/minute
Arm/Group | CSJ117 0.5mg | CSJ117 1mg | CSJ117 2mg | CSJ117 4mg | CSJ117 8mg | Placebo
Number analyzed (Participants) | 31 | 33 | 32 | 65 | 66 | 61
liters/minute | -0.9785 (22.73169) | -1.7035 (28.83957) | 18.9496 (50.09045) | -0.0319 (33.56218) | 3.5702 (37.05293) | -2.2060 (24.56187)

4. Secondary Outcome: Change From Baseline in Evening PEF at Week 12
Description: as for outcome 3
Time Frame: Baseline, Week 12
Population: Participants in the Full Analysis Set with a valid measurement for the outcome measure
Measure: Mean (Standard Deviation); unit: liters/minute
Arm/Group | CSJ117 0.5mg | CSJ117 1mg | CSJ117 2mg | CSJ117 4mg | CSJ117 8mg | Placebo
Number analyzed (Participants) | 29 | 30 | 31 | 59 | 62 | 58
liters/minute | -5.3894 (29.13968) | -7.8709 (29.06055) | 14.0265 (44.90062) | 0.3893 (30.47064) | 2.6905 (32.27860) | -3.2785 (22.93816)

5. Secondary Outcome: Average Change From Baseline in ACQ-5 Score at Week 8 and Week 12
Description: The Asthma Control Questionnaire-5 (ACQ-5) is a five-item, self-completed questionnaire, which is used as a measure of asthma symptom control. Patients were asked to recall how their asthma had been during the previous week and to respond to the symptom questions on a 7-point scale (0=no impairment, 6=maximum impairment). The questions are equally weighted and the overall ACQ-5 score is the mean of all 5 questions, therefore between 0 (totally controlled) and 6 (severely uncontrolled).
  The baseline values of ACQ-5 were collected at the end of the run-in period. The least-squares means for change from baseline in ACQ-5 score averaged between Week 8 and Week 12 visits for each individual dose group were obtained from a linear mixed effects model for repeated measures (MMRM).
  A negative change from baseline in ACQ-5 is considered a favorable outcome.
Time Frame: Baseline, Weeks 8-12
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CSJ117 0.5mg | CSJ117 1mg | CSJ117 2mg | CSJ117 4mg | CSJ117 8mg | Placebo
Number analyzed (Participants) | 36 | 37 | 37 | 76 | 74 | 75
score on a scale | -0.764 (0.1230) | -1.142 (0.1225) | -1.011 (0.1171) | -0.739 (0.0824) | -0.837 (0.0829) | -0.722 (0.0846)
Statistical Analysis 1: Comparison: CSJ117 0.5mg vs Placebo; Test type: Superiority; p = 0.780, MMRM; Least Squares mean = -0.042, 95% CI 2-sided [-0.336 to 0.252], Standard Error of Mean 0.1493 — Treatment difference (CSJ117-placebo)
Statistical Analysis 2: Comparison: CSJ117 1mg vs Placebo; Test type: Superiority; p = 0.005, MMRM; Least Squares mean = -0.420, 95% CI 2-sided [-0.713 to -0.127], Standard Error of Mean 0.1489 — Treatment difference (CCSJ117-placebo)
Statistical Analysis 3: Comparison: CSJ117 2mg vs Placebo; Test type: Superiority; p = 0.047, MMRM; Least Squares mean = -0.289, 95% CI 2-sided [-0.573 to 0.004], Standard Error of Mean 0.1446 — Treatment difference (CCSJ117-placebo)
Statistical Analysis 4: Comparison: CSJ117 4mg vs Placebo; Test type: Superiority; p = 0.887, MMRM; Least Squares mean = -0.017, 95% CI 2-sided [-0.249 to 0.216], Standard Error of Mean 0.1182 — Treatment difference (CCSJ117-placebo)
Statistical Analysis 5: Comparison: CSJ117 8mg vs Placebo; Test type: Superiority; p = 0.333, MMRM; Least Squares mean = -0.115, 95% CI 2-sided [-0.348 to 0.118], Standard Error of Mean 0.1184 — Treatment difference (CCSJ117-placebo)

6. Secondary Outcome: Average Change From Baseline in AQLQ+12 Score at Week 8 and Week 12
Description: The Asthma Quality of Life Questionnaire+12 (AQLQ+12) is a disease specific questionnaire, which is used as a measure of health-related quality of life. The AQLQ+12 comprises a total of 32 individual questions that span a total of 4 domains: symptoms, activity limitation, emotional function, and environmental stimuli. Patients are asked to recall their experiences during the previous 2 weeks and to score each item on a 7-point scale (7 = not at all impaired to 1 = severely impaired). The overall AQLQ+12 score is the mean of all 32 individual responses, therefore between 7 and 1 with higher scores indicating less impairment in health-related quality of life.
  The baseline values of AQLQ+12 were collected at the end of the run-in period. The least-squares means for change from baseline in AQLQ+12 score averaged between Week 8 and Week 12 visits were obtained from a linear mixed effects model for repeated measures (MMRM).
  A positive change from baseline is considered a favorable outcome.
Time Frame: Baseline, Weeks 8-12
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | CSJ117 0.5mg | CSJ117 1mg | CSJ117 2mg | CSJ117 4mg | CSJ117 8mg | Placebo
Number analyzed (Participants) | 36 | 37 | 37 | 76 | 74 | 75
score on a scale | 0.467 (0.1223) | 0.781 (0.1220) | 0.642 (0.1177) | 0.597 (0.0828) | 0.636 (0.0826) | 0.564 (0.0842)
Statistical Analysis 1: Comparison: CSJ117 0.5mg vs Placebo; Test type: Superiority; p = 0.515, MMRM; Least Squares mean = -0.097, 95% CI 2-sided [-0.389 to 0.195], Standard Error of Mean 0.1485 — Treatment difference (CSJ117-placebo)
Statistical Analysis 2: Comparison: CSJ117 1mg vs Placebo; Test type: Superiority; p = 0.143, MMRM; Least Squares mean = 0.218, 95% CI 2-sided [-0.074 to 0.510], Standard Error of Mean 0.1484 — Treatment difference (CCSJ117-placebo)
Statistical Analysis 3: Comparison: CSJ117 2mg vs Placebo; Test type: Superiority; p = 0.590, MMRM; Least Squares mean = 0.078, 95% CI 2-sided [-0.207 to 0.364], Standard Error of Mean 0.1450 — Treatment difference (CCSJ117-placebo)
Statistical Analysis 4: Comparison: CSJ117 4mg vs Placebo; Test type: Superiority; p = 0.778, MMRM; Least Squares mean = 0.033, 95% CI 2-sided [-0.199 to 0.265], Standard Error of Mean 0.1180 — Treatment difference (CCSJ117-placebo)
Statistical Analysis 5: Comparison: CSJ117 8mg vs Placebo; Test type: Superiority; p = 0.539, MMRM; Least Squares mean = 0.073, 95% CI 2-sided [-0.160 to 0.305], Standard Error of Mean 0.1180 — Treatment difference (CCSJ117-placebo)

7. Secondary Outcome: Change From Baseline in ADSD Score at Week 8 and Week 12
Description: Asthma Daytime Symptom Diary (ADSD) and Asthma Nighttime Symptom Diary (ANSD) are patient reported outcome measures of asthma symptom severity.
  Patients recorded asthma symptoms twice daily in the eDiary. Severity of daytime asthma symptoms were assessed before going to bed and severity of nighttime symptoms upon waking.
  Both diaries comprised of 6 items assessing breathing symptoms (difficulty breathing, wheezing, and shortness of breath), chest symptoms (chest tightness and chest pain), and cough symptoms (cough). All items were assessed using an 11-point numeric rating scale ranging from 0 ('None') to 10 ('As bad as you can imagine'). The overall score is the mean of all 6 individual responses, therefore between 0 and 10 with higher scores indicating more severe symptoms.
  Mean daily scores of both diaries were calculated by weekly intervals. The baseline values were defined as the average score during the run-in period.
  A negative change from baseline is a favorable outcome.
Time Frame: Baseline, Week 8 and Week 12
Population: Participants in the Full Analysis Set with a valid measurement for the outcome measure at each timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CSJ117 0.5mg | CSJ117 1mg | CSJ117 2mg | CSJ117 4mg | CSJ117 8mg | Placebo
Number analyzed (Participants) | 33 | 33 | 37 | 73 | 72 | 67
score on a scale
  Week 8 | -0.24 (0.678) | -0.42 (0.622) | -0.35 (0.773) | -0.32 (0.555) | -0.33 (0.787) | -0.25 (0.580)
  Week 12: number analyzed (Participants) | 32 | 32 | 32 | 68 | 65 | 64
  Week 12 | -0.29 (0.752) | -0.59 (0.938) | -0.38 (0.687) | -0.33 (0.581) | -0.35 (0.820) | -0.37 (0.754)

8. Secondary Outcome: Change From Baseline in ANSD Score at Week 8 and Week 12
Description: as for outcome 7
Time Frame: Baseline, Week 8 and Week 12
Population: Participants in the Full Analysis Set with a valid measurement for the outcome measure at each timepoint
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CSJ117 0.5mg | CSJ117 1mg | CSJ117 2mg | CSJ117 4mg | CSJ117 8mg | Placebo
Number analyzed (Participants) | 34 | 34 | 37 | 74 | 72 | 69
score on a scale
  Week 8: number analyzed (Participants) | 33 | 34 | 37 | 74 | 72 | 69
  Week 8 | -0.15 (0.637) | -0.35 (0.629) | -0.30 (0.760) | -0.27 (0.547) | -0.26 (0.753) | -0.25 (0.634)
  Week 12: number analyzed (Participants) | 34 | 33 | 35 | 70 | 69 | 66
  Week 12 | -0.19 (0.480) | -0.46 (0.868) | -0.29 (0.695) | -0.26 (0.590) | -0.23 (0.769) | -0.33 (0.729)

9. Secondary Outcome: Change From Baseline in Number of Puffs of SABA Taken Per Day at Week 12
Description: Participants were given a short acting β2-agonist (SABA) such as salbutamol (100 µg) or albuterol (90 µg) to use as rescue medication throughout the study. Participants recorded in the eDiary, once in the morning and once in the evening, the use of rescue medication (number of puffs of SABA taken in the previous 12 hours). The total number of puffs of SABA taken per day was calculated and the mean daily use of puffs of SABA was derived by weekly intervals.
  The baseline value of number of puffs of SABA taken per day is the average of total daily SABA use during the run-in period.
  A negative change from baseline is considered a favorable outcome.
Time Frame: Baseline, Week 12
Population: Participants in the Full Analysis Set with a valid measurement for the outcome measure
Measure: Mean (Standard Deviation); unit: puffs of SABA per day
Arm/Group | CSJ117 0.5mg | CSJ117 1mg | CSJ117 2mg | CSJ117 4mg | CSJ117 8mg | Placebo
Number analyzed (Participants) | 34 | 33 | 35 | 70 | 70 | 68
puffs of SABA per day | -0.2189 (0.72340) | -0.4548 (0.88125) | -0.3420 (0.68267) | -0.4310 (0.80279) | -0.3766 (0.98070) | -0.3543 (0.78420)

10. Secondary Outcome: Number of Participants With On-treatment Adverse Events (AEs) and Serious Adverse Events (SAEs) During the On-treatment Period
Description: Number of participants with AEs and SAEs, including asthma exacerbations, changes from baseline in vital signs, electrocardiograms and laboratory results qualifying and reported as AEs during the on-treatment period.
  The on-treatment period is between the date of first dose of double-blind study treatment and date of the last dose of randomized study treatment.
  Grades to characterize the severity of the adverse events were based on the Common Terminology Criteria for Adverse Events (CTCAE). For CTCAE, Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening; Grade 5 = death related to AE.
  The number of participants in each category is reported in the table.
Time Frame: From first dose of double-blind study treatment up to last dose (Week 12)
Population: Safety Analysis Set defined as participants who received at least one dose of double-blind treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | CSJ117 0.5mg | CSJ117 1mg | CSJ117 2mg | CSJ117 4mg | CSJ117 8mg | Placebo
Number analyzed (Participants) | 36 | 37 | 37 | 76 | 74 | 75
Participants
  At least one AE | 12 | 10 | 13 | 22 | 25 | 23
  Mild AEs | 5 | 8 | 6 | 9 | 13 | 13
  Moderate AEs | 6 | 2 | 7 | 12 | 12 | 10
  Severe AEs | 1 | 0 | 0 | 1 | 0 | 0
  Study treatment-related AEs | 0 | 1 | 1 | 2 | 4 | 2
  SAEs | 1 | 0 | 0 | 0 | 0 | 1
  AEs leading to discontinuation | 1 | 0 | 0 | 0 | 0 | 2

11. Secondary Outcome: Number of Participants With Anti-CSJ117 Antibodies
Description: Immunogenicity (antibody formation against CSJ117) was evaluated in serum by a validated bridging electrochemiluminescence immunoassay (ECLIA).
Time Frame: Day 1 and Weeks 2, 4, 8, 12, 14, 16, 20 and 24
Population: Participants in the Safety Analysis Set with a valid measurement for the outcome measure. Safety Analysis Set is defined as participants who received at least one dose of double-blind treatment. The number analyzed per row represents participants with data at the corresponding time point.
Measure: Count of Participants; unit: Participants
Arm/Group | CSJ117 0.5mg | CSJ117 1mg | CSJ117 2mg | CSJ117 4mg | CSJ117 8mg | Placebo
Number analyzed (Participants) | 36 | 36 | 37 | 76 | 74 | 75
Participants
  Day 1: Negative | 30 | 33 | 31 | 66 | 63 | 63
  Day 1: Positive | 6 | 3 | 6 | 10 | 11 | 12
  Week 2: number analyzed (Participants) | 35 | 35 | 37 | 75 | 74 | 69
  Week 2: Negative | 27 | 31 | 31 | 65 | 64 | 56
  Week 2: Positive | 8 | 4 | 6 | 10 | 10 | 13
  Week 4: number analyzed (Participants) | 33 | 35 | 37 | 74 | 71 | 71
  Week 4: Negative | 26 | 29 | 26 | 49 | 47 | 57
  Week 4: Positive | 7 | 6 | 11 | 25 | 24 | 14
  Week 8: number analyzed (Participants) | 34 | 33 | 37 | 72 | 72 | 67
  Week 8: Negative | 17 | 16 | 10 | 22 | 18 | 58
  Week 8: Positive | 17 | 17 | 27 | 50 | 54 | 9
  Week 12: number analyzed (Participants) | 33 | 33 | 35 | 71 | 71 | 66
  Week 12: Negative | 9 | 11 | 5 | 19 | 11 | 53
  Week 12: Positive | 24 | 22 | 30 | 52 | 60 | 13
  Week 14: number analyzed (Participants) | 26 | 25 | 29 | 59 | 52 | 56
  Week 14: Negative | 7 | 6 | 3 | 13 | 6 | 49
  Week 14: Positive | 19 | 19 | 26 | 46 | 46 | 7
  Week 16: number analyzed (Participants) | 26 | 25 | 29 | 58 | 53 | 56
  Week 16: Negative | 7 | 8 | 3 | 12 | 7 | 49
  Week 16: Positive | 19 | 17 | 26 | 46 | 46 | 7
  Week 20: number analyzed (Participants) | 26 | 25 | 29 | 58 | 53 | 55
  Week 20: Negative | 9 | 9 | 6 | 13 | 6 | 47
  Week 20: Positive | 17 | 16 | 23 | 45 | 47 | 8
  Week 24: number analyzed (Participants) | 26 | 25 | 28 | 56 | 53 | 56
  Week 24: Negative | 11 | 10 | 5 | 13 | 8 | 49
  Week 24: Positive | 15 | 15 | 23 | 43 | 45 | 7

12. Secondary Outcome: CSJ117 Serum Concentration
Description: CSJ117 concentration was determined in serum by a validated immunoassay method. Concentrations below the lower limit of quantification (LLOQ) were treated as "zero".
Time Frame: Day 1 and Week 12: pre-dose, 2 and 4 hours post-dose; Weeks 2, 4 and 8: pre-dose and 4 hours post-dose; Weeks 14, 16, 20 and 24: pre-dose
Population: Participants in the PK set with a valid measurement for the outcome measure. PK set is defined as participants with at least one evaluable drug concentration data sample. The number analyzed per row represents participants with data at the corresponding time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CSJ117 0.5mg | CSJ117 1mg | CSJ117 2mg | CSJ117 4mg | CSJ117 8mg
Number analyzed (Participants) | 36 | 37 | 37 | 75 | 74
ng/mL
  Day 1, pre-dose: number analyzed (Participants) | 36 | 37 | 36 | 74 | 73
  Day 1, pre-dose | 0.00 (0.00) | 0.00 (0.00) | 1.34 (8.02) | 0.00 (0.00) | 0.00 (0.00)
  Day 1, 2 hours post-dose: number analyzed (Participants) | 36 | 37 | 37 | 74 | 74
  Day 1, 2 hours post-dose | 0.00 (0.00) | 0.00 (0.00) | 1.86 (7.36) | 0.00 (0.00) | 0.157 (0.947)
  Day 1, 4 hours post-dose: number analyzed (Participants) | 36 | 37 | 37 | 74 | 73
  Day 1, 4 hours post-dose | 0.00 (0.00) | 0.00 (0.00) | 1.97 (7.90) | 0.214 (1.33) | 0.924 (2.58)
  Week 2, pre-dose: number analyzed (Participants) | 35 | 35 | 37 | 75 | 74
  Week 2, pre-dose | 0.320 (1.89) | 0.00 (0.00) | 2.32 (8.57) | 2.00 (4.74) | 6.58 (7.61)
  Week 2, 2 hours post-dose: number analyzed (Participants) | 35 | 34 | 37 | 73 | 74
  Week 2, 2 hours post-dose | 0.389 (2.30) | 0.00 (0.00) | 2.20 (8.05) | 1.66 (3.51) | 7.66 (7.83)
  Week 4, pre-dose: number analyzed (Participants) | 33 | 35 | 36 | 74 | 70
  Week 4, pre-dose | 0.336 (1.93) | 0.00 (0.00) | 2.89 (9.03) | 2.86 (5.11) | 12.0 (19.5)
  Week 4, 2 hours post-dose: number analyzed (Participants) | 33 | 34 | 37 | 74 | 69
  Week 4, 2 hours post-dose | 0.467 (2.68) | 0.00 (0.00) | 3.19 (9.01) | 3.59 (5.69) | 13.8 (22.2)
  Week 8, pre-dose: number analyzed (Participants) | 33 | 33 | 37 | 72 | 71
  Week 8, pre-dose | 1.69 (4.34) | 3.15 (6.50) | 6.79 (12.0) | 11.5 (15.8) | 39.3 (51.0)
  Week 8, 2 hours post-dose: number analyzed (Participants) | 33 | 33 | 36 | 71 | 68
  Week 8, 2 hours post-dose | 1.84 (4.69) | 3.29 (6.85) | 6.94 (12.2) | 11.1 (14.7) | 39.8 (49.9)
  Week 12, pre-dose: number analyzed (Participants) | 32 | 33 | 31 | 69 | 70
  Week 12, pre-dose | 1.83 (4.69) | 2.20 (4.61) | 10.3 (16.8) | 14.6 (20.3) | 49.5 (62.1)
  Week 12, 2 hours post-dose: number analyzed (Participants) | 32 | 32 | 31 | 68 | 68
  Week 12, 2 hours post-dose | 2.02 (4.68) | 2.49 (4.81) | 10.2 (16.4) | 14.3 (20.3) | 45.7 (49.7)
  Week 12, 4 hours post-dose: number analyzed (Participants) | 32 | 32 | 31 | 68 | 68
  Week 12, 4 hours post-dose | 2.11 (4.84) | 2.51 (4.79) | 10.1 (16.3) | 15.2 (20.7) | 46.7 (52.2)
  Week 14, pre-dose: number analyzed (Participants) | 25 | 25 | 27 | 58 | 52
  Week 14, pre-dose | 0.239 (1.19) | 0.00 (0.00) | 2.97 (10.1) | 1.59 (4.43) | 7.26 (15.7)
  Week 16, pre-dose: number analyzed (Participants) | 25 | 25 | 27 | 57 | 53
  Week 16, pre-dose | 0.00 (0.00) | 0.00 (0.00) | 2.16 (10.0) | 0.424 (1.92) | 2.53 (8.10)
  Week 20, pre-dose: number analyzed (Participants) | 25 | 25 | 27 | 58 | 53
  Week 20, pre-dose | 0.00 (0.00) | 0.00 (0.00) | 1.94 (8.99) | 0.00 (0.00) | 0.163 (1.19)
  Week 24, pre-dose: number analyzed (Participants) | 25 | 25 | 26 | 55 | 53
  Week 24, pre-dose | 0.00 (0.00) | 0.00 (0.00) | 1.86 (6.81) | 0.00 (0.00) | 0.00 (0.00)

ADVERSE EVENTS:
Time Frame: From first dose of double-blind study treatment up to 12 weeks after last dose (Week 24)
Groups:
- CSJ117 8mg: CSJ117 1 mg inhaled once daily
Arm/Group | CSJ117 0.5mg | CSJ117 1mg | CSJ117 2mg | CSJ117 4mg | CSJ117 8mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/37 | 0/37 | 0/76 | 0/74 | 0/75
Serious Adverse Events (participants affected / at risk) | 1/36 | 0/37 | 0/37 | 1/76 | 0/74 | 1/75
Other Adverse Events (participants affected / at risk) | 12/36 | 14/37 | 20/37 | 31/76 | 23/74 | 27/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CSJ117 0.5mg (N=36) | CSJ117 1mg (N=37) | CSJ117 2mg (N=37) | CSJ117 4mg (N=76) | CSJ117 8mg (N=74) | Placebo (N=75)
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CSJ117 0.5mg (N=36) | CSJ117 1mg (N=37) | CSJ117 2mg (N=37) | CSJ117 4mg (N=76) | CSJ117 8mg (N=74) | Placebo (N=75)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Vaccination site swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 1 | 1 | 0
COVID-19 (Infections and infestations) | 4 | 2 | 0 | 3 | 1 | 7
Candida infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 3 | 3 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 2 | 1 | 4 | 2 | 4
Oral fungal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Papilloma viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 2 | 2 | 2
Pharyngitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 2 | 1 | 3 | 2
Tracheitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 2 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 1 | 0 | 1
Blood glucose increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 1 | 2
Migraine (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Spinal cord herniation (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 6 | 12 | 7 | 10
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chronic rhinosinusitis with nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 3 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0 | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-01-21): https://cdn.clinicaltrials.gov/large-docs/23/NCT04410523/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-22): https://cdn.clinicaltrials.gov/large-docs/23/NCT04410523/SAP_001.pdf